CLINICAL TRIAL: NCT06570915
Title: A Prospective, Single-arm, Multicenter, Open-label , Phase 2 Study to Evaluate Efficacy and Safety of the Daratumumab in T Cell Acute Lymphoblastic Leukemia With Minimal Residual-Positive After Standard Chemotherapy
Brief Title: Daratumumab for T Cell ALL With MRD-positive After Standard Chemotherapy
Acronym: T-ALL-2024
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024056
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: ALL, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab (Experimental): Daratumumab was administered once a week at a dose of 16 mg/kg for a total of 4 times (Day1,8,15,22 dosing patterns) in one cycle. Patients with conditions may use up to two cycles of treatment.
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — Daratumumab was administered once a week at a dose of 16 mg/kg for a total of 4 times (Day1,8,15,22 ) in one cycle.

SUMMARY:
T-ALL accounts for about 15%-25% of Ph-negative ALL, and its clinical prognosis is worse than B-ALL. The successful application of immunotherapy has brought revolutionary progress to the treatment of ALL. But progress in the treatment of T-ALL has been relatively slow. Minimal residual disease (MRD) is a strong prognostic indicator for ALL patients. MRD-positive after induction therapy predicts a high risk of relapse. The National Comprehensive Cancer Network (NCCN) considers MRD-positive ALL patients to be at high risk. Research in the B-ALL field has demonstrated that immunotherapy has the potential to further clear MRD, which in turn translates into survival benefits. Daratumumab is a humanized, anti-CD38 IgG1 monoclonal antibody that binds to CD38 expressed by tumor cells. Apoptosis of tumor cells is induced through a variety of immune-related mechanisms such as complement-dependent cytotoxicity (CDC), antibody-dependent cell-mediated cytotoxicity (ADCC), antibody-dependent cytophagocytosis (ADCP), and FCγ receptors, which are currently mainly used in the treatment of multiple myeloma. CD38 is highly and stably expressed on the surface of T-ALL cells, and its expression was less influenced by the previous treatment. Preliminary data from the clinical study of daratumumab combined with BFM bone frame prescription for the treatment of recurrent refractory T ALL(NCT03384654) showed that the effectiveness rate (ORR) was 83.3% in children and 60% in young adults. Compared with the previous historical data, the safety and tolerability were significantly improved. For T-ALL patients who relapse after allogeneic transplantation and achieve CR with intense chemotherapy but continue to have MRD-positive flow rate, daratumumab monotherapy can further clear MRD and achieve the purpose of sustaining CR. These studies all demonstrate the potential role of daratumumab in the treatment of T-ALL. Based on the current difficulties in the treatment of T-ALL and existing research data, we plan to conduct a prospective, single-arm, open-label phase II clinical study to explore the efficacy and safety of daratumumab for flow minimal residual disease positive T-ALL after standard chemotherapy.

DETAILED DESCRIPTION:
Daratumumab is administered once a week at a dose of 16 mg/kg for a total of 4 times (Day1,8,15,22) in one cycle. Conditions patients can use up to two cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed T-cell acute lymphoblastic leukemia confirmed by cell morphology and immunophenotype had flow MRD≥0.01% 3 months after chemotherapy; or patients with T-cell acute lymphoblastic leukemia relapsed achieved CR again after salvage chemotherapy, but the flow MRD was ≥0.01%
2. Age ≥18 years old, male or female
3. The expression of CD38 in tumor cells was positive
4. Men and women who may give birth agree to and use effective contraceptive methods
5. Main organ function assessment criteria: total bilirubin < 1.5× upper normal limit (ULN), glutamic oxalic aminotransferase (AST) and glutamic alanine aminotransferase (ALT) ≤2.5×ULN; Serum creatinine < 2×ULN; Myocardial enzyme < 2×ULN; Serum amylase ≤1.5×ULN; Left ventricular ejection fraction (LEF) was > 45%
6. Understand and sign the informed consent and agree to comply with the study requirements

Exclusion Criteria:

1. SAEs related to the study emerged during the study, and the investigator judged that the necessity of quitting the project was greater than the benefit
2. In case of any situation in which the subjects could not tolerate the study regimen, the investigator assessed that the necessity of withdrawal from the regimen outweighed the benefit
3. The subject had an allergic reaction to any drug of the study regimen or other conditions that prevented the regimen from continuing
4. Subjects voluntarily asked to withdraw from the study at any time
5. Any situation in which the investigator determines that the benefit of withdrawing from the study outweighs the benefit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion from MRD+to MRD- by flow cytometry after 1 cycle of daretuzumab treatment | up to 28days ±3days after daretuzumab treatment
  If no abnormal phenotypic leukemia cells were detected by flow cytometry, flow MRD-negative was considered

SECONDARY OUTCOMES:
overall survival overall survival overall survival | up to 2 years after the date of the last enrolled participants
  The interval from the date of enrollment to the date of death or the date of last follow-up, whichever occurred first.
Disease-free survival (DFS) | up to 2 years after the date of the last enrolled participants
  Only for CR patients who chieved CR. The interval from the date of CR1 to relapse, death from any cause or last follow-up.
Cumulative incidence of relapse (CIR) | up to 2 years after the date of the last enrolled participants
  Calculated with the cumulative incidence method, with death in patients who had a complete hematologic response as a competing risk.
duration of MRD-negative response | up to 2 years after the date of the last enrolled participants
  No blasts were detected by flow cytometry after daretuzumab treatment
Rate of conversion from MRD+to MRD- by NGS | up to 2 years after the date of the last enrolled participants
  Next-generation sequencing (NGS) is a high-throughput sequencing methodology and is a process by which small fragments of DNA are sequenced in parallel multiple times
30-day mortality | Within 30 days of the date of the last enrolled participants
  Percentage of patients who died within 30 days from enrollment
60-day mortality | Within 60 days of the date of the last enrolled participants
  Percentage of patients who died within 60 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, doctor, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College

IPD SHARING:
Plan to Share IPD: No